CLINICAL TRIAL: NCT02684097
Title: A Randomized Placebo-controlled Single Center Pilot Study of the Safety and Efficacy of Tralokinumab in Subjects With Moderate to Severe Alopecia Areata
Brief Title: A Pilot Study of Tralokinumab in Subjects With Moderate to Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emma Guttman (Other)
Responsible Party: Sponsor-Investigator, Emma Guttman, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 15-1497
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Alopecia Areata
Keywords: Alopecia, Alopecia Totalis, Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tralokinumab (Active Comparator): Tralokinumab subcutaneous injection every two weeks for 24 weeks
  Interventions: Drug: Tralokinumab
- Placebo (Placebo Comparator): Saline subcutaneous injection every two weeks for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tralokinumab — All groups will receive study drug every two weeks for 24 weeks.
  Arms: Tralokinumab
Drug: Placebo — Matching placebo given every two weeks for 24 weeks
  Other Names: Saline subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether tralokinumab can be a helpful treatment for alopecia areata. This is a randomized, double-blind, placebo-controlled pilot study of a total of 30 subjects with moderate to severe alopecia areata involving 30-100% of the scalp. Expected is 50% of these subjects to have concomitant alopecia areata (AA) and atopic dermatitis (AD). Subjects with AA alone (15 subjects) will be randomized (2:1) to either receive tralokinumab or placebo via subcutaneous injection every 2 weeks for 24 weeks. Subjects with concomitant alopecia areata and atopic dermatitis (15 subjects) will be randomized separately in a 2:1 ratio to receive tralokinumab or placebo via subcutaneous injection every 2 weeks for 24 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether tralokinumab can be a helpful treatment for alopecia areata.

This is a randomized, double-blind, placebo-controlled pilot study of a total of 30 subjects with moderate to severe alopecia areata involving 30-100% of the scalp. The researchers expect 50% of these subjects to have concomitant alopecia areata (AA) and atopic dermatitis (AD).

The researchers' experience in AD12-14, and past experience in psoriasis15, 16 showed that biomarker studies in skin tissues are critical to the understanding of key pathogenic pathways that are upregulated in each disease and how well they are suppressed with effective treatment. These mechanistic studies coupled with clinical trials are key in the disease to shed light on important disease mechanisms, and to explain which molecules are suppressed by each therapeutic target. Data shows that IL-13 is significantly upregulated in both AD and AA lesions compared to nonlesional skin. It is very important to associate the clinical responses with suppression of this cytokine and related molecules as well as other pathway cytokines in skin tissues. Both the whole genomic profiling and individual molecular and cellular markers are very important in order to understand how well anti-IL-13 will change/suppress AA-associated pathways and compare with those that will be suppressed in AD.

Since this study is designed to gain basic knowledge rather than to yield information directly related to patient care, the results are not entered in the participants' medical records. If, at a later date, correlations of in-vitro tests and the patients' clinical situation suggest that the results do bear on the patients' health, an amended protocol will be submitted to the IRB so that results can be made available to the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18 to 75 years, inclusively at the time of signing the informed consent document.
* Subject has provided written informed consent prior to any study specific procedures.
* Body weight of ≥40 and <150 kg at enrollment.
* Subject has a history of alopecia areata for at least 3 months.
* Subject has extensive patchy alopecia areata (at least 30% scalp hair loss).
* No evidence of hair regrowth at Baseline.
* For WOCBP only: have a negative urine pregnancy test prior to administration of the IP.
* For inclusion in the voluntary pharmacogenetic research, subjects should fulfill the following criterion: Provision of a signed and dated written informed consent for the pharmacogenetic sample and analysis. If a subject declines to participate in the pharmacogenetic research, there will be no consequence or loss of benefit to the subject. The subject will not be excluded from the other aspects of the study described in the protocol, as long as they consent to participate in the study.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination performed at Screening.
* Subjects may be naïve to treatment or unresponsive to intralesional steroids or other treatments for alopecia areata.

Exclusion Criteria:

* History of male or female pattern hair loss Ludwig stage III or Hamilton > stage V.
* Subjects in whom the diagnosis of alopecia areata is in question.
* Any disorder, including but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

  1. Affect the safety of the subject throughout the study
  2. Influence the findings of the studies or their interpretations
  3. Impede the subject's ability to complete the entire duration of study
* Known history of allergy or reaction to any component of the IP formulation.
* History of anaphylaxis following any biologic therapy.
* The following treatments within 4 weeks before the Baseline visit, or any condition that, in the opinion of the investigator, will likely require such treatment(s) at any time during the study:

  1. Systemic corticosteroids
  2. Immunosuppressive/immunomodulating drugs (eg, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase (JAK) inhibitors, azathioprine or methotrexate), Ultra-Violet (UV) B phototherapy; and/or Psoralen Ultra-Violet A (PUVA) therapy.
* Treatment with topical corticosteroids, tacrolimus and/or pimecrolimus within 1 week before the Baseline visit.
* Subject has taken enzyme-modifying drugs that are moderate inhibitors/potent inducers of cytochrome P450 3A4 or potent inhibitors of cytochrome P450 2C19 enzymes (such as cimetidine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole etc…) and strong inducers of CYP enzymes (such as rifampin etc…), in the previous 28 days before day 0.
* A helminth parasitic infection diagnosed within 6 months prior to the date informed consent or assent obtained that has not been treated with, or has failed to respond to, standard of care therapy.
* History of clinically significant infection, including acute upper or lower respiratory infections, requiring antibiotics or antiviral medication within 30 days prior to the date informed consent or assent is obtained or during the run-in period.
* Tuberculosis requiring treatment within the 12 months prior to enrolment (Visit 1).
* Any clinically significant abnormal findings in physical examination, vital signs, ECG, hematology, clinical chemistry, or urinalysis during the run-in period, which in the opinion of the Investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to complete entire duration of the study.
* History of chronic alcohol or drug abuse within 12 months of the enrolment visit, or a condition associated with poor compliance as judged by the Investigator.
* Positive hepatitis B surface antigen or hepatitis C virus antibody serology. Subjects with a history of hepatitis B vaccination without a history of hepatitis B are allowed to be enrolled.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at enrolment, or the subject taking antiretroviral medications as determined by medical history and/or subject's verbal report.
* Current tobacco smoking (smoking must have stopped for ≥ 3 months prior to enrollment) or a history of tobacco smoking for ≥ 10 pack-years (one pack year = 20 cigarettes smoked per day for 1 year).
* History of cancer: - Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained
* Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, systemic corticosteroids including regular treatment with OCS or intramuscular long-acting depot corticosteroids, or any experimental anti-inflammatory therapy) within 3 months prior to the date informed consent or assent is obtained.
* Clinically significant asthma exacerbation, in the opinion of the Investigator, including those requiring use of oral corticosteroids 30 days prior to the date of informed consent or during the screening/run-in period.
* Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent or assent is obtained.
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives prior to the enrolment visit, whichever is longer.
* Receipt of live attenuated vaccines 30 days prior to the date of randomization and during the study including the follow-up period Receipt of inactive/killed vaccinations (eg, inactive influenza) are allowed, provided they are not administered within 5 days before/after any study visit.
* Receipt of any investigational non-biologic agent within 30 days or 5 half lives prior to informed consent or assent being obtained, whichever is longer.
* Previous receipt of tralokinumab (CAT-354).
* Initiation of new allergen immunotherapy or change in existing immunotherapy is not allowed within 30 days prior to the date of informed consent. However allergen immunotherapy initiated prior to this period may be continued provided there is a span of at least 5 days between the immunotherapy and IP administration.
* Current use of oral or ophthalmic non-selective β-adrenergic antagonist (eg, propranolol).
* Current use of five- lipoxygenase inhibitors (eg, Zileuton) or roflumilast.
* Major surgery within 8 weeks prior to the enrolment visit, or planned in-subject surgery or hospitalization during the study period.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.5 times the upper limit of normal (ULN) at enrolment
* Pregnant, currently breast-feeding, or lactating women.
* Previous randomization in the present study.
* Concurrent enrollment in another clinical study where the subject is receiving an IP.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Employees of the clinical study site or any other individuals directly involved with the planning or conduct of the study, or immediate family members of such individuals.
* Individuals who are legally institutionalized.

For exclusion from the voluntary pharmacogenetic research:

* Previous allogeneic bone marrow transplant.
* Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — ISMMS
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkhalifah A. Alopecia areata update. Dermatol Clin. 2013 Jan;31(1):93-108. doi: 10.1016/j.det.2012.08.010. Epub 2012 Oct 2. PMID 23159179
- [Background] Safavi KH, Muller SA, Suman VJ, Moshell AN, Melton LJ 3rd. Incidence of alopecia areata in Olmsted County, Minnesota, 1975 through 1989. Mayo Clin Proc. 1995 Jul;70(7):628-33. doi: 10.4065/70.7.628. PMID 7791384
- [Background] Huang KP, Mullangi S, Guo Y, Qureshi AA. Autoimmune, atopic, and mental health comorbid conditions associated with alopecia areata in the United States. JAMA Dermatol. 2013 Jul;149(7):789-94. doi: 10.1001/jamadermatol.2013.3049. PMID 23700152
- [Background] Betz RC, Pforr J, Flaquer A, Redler S, Hanneken S, Eigelshoven S, Kortum AK, Tuting T, Lambert J, De Weert J, Hillmer AM, Schmael C, Wienker TF, Kruse R, Lutz G, Blaumeiser B, Nothen MM. Loss-of-function mutations in the filaggrin gene and alopecia areata: strong risk factor for a severe course of disease in patients comorbid for atopic disease. J Invest Dermatol. 2007 Nov;127(11):2539-43. doi: 10.1038/sj.jid.5700915. Epub 2007 Jun 21. PMID 17581619
- [Background] Olsen EA, Hordinsky MK, Price VH, Roberts JL, Shapiro J, Canfield D, Duvic M, King LE Jr, McMichael AJ, Randall VA, Turner ML, Sperling L, Whiting DA, Norris D; National Alopecia Areata Foundation. Alopecia areata investigational assessment guidelines--Part II. National Alopecia Areata Foundation. J Am Acad Dermatol. 2004 Sep;51(3):440-7. doi: 10.1016/j.jaad.2003.09.032. No abstract available. PMID 15337988

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tralokinumab | Placebo
Started | 15 | 7
Completed | 2 | 1
Not Completed | 13 | 6
Not completed — Lack of Efficacy | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab | Placebo | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.67 (12.45) | 47.57 (16.37) | 44.23 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Severity of Alopecia Tool (SALT) [Mean (Standard Deviation); unit: units on a scale] — SALT score 0-100 with lower score indicating better health outcomes
  units on a scale | 80.92 (25.65) | 72.25 (25.51) | 78.16 (25.33)
Alopecia Areata Symptom Impact Scale (AASIS) [Mean (Standard Deviation); unit: units on a scale] — AASIS score 0-130 with lower score indicating better health outcomes
  units on a scale | 54.67 (28.04) | 51.57 (21.19) | 53.68 (25.59)
Alopecia Areata Quality of Life (AA-QoL) [Mean (Standard Deviation); unit: units on a scale] — AA-QoL score 0-100 with higher score indicating better health outcomes
  units on a scale | 51.07 (12.98) | 51.57 (7.82) | 51.23 (11.39)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gene Expression Th2/IL-13, "T22"/IL-22, S100A7 and S100A8, Th1/IFN-gamma, and Th17/IL-17A Jointly Correlated
Description: Change from baseline in cellular, and molecular markers in skin biopsies after treatment. Gene expression changes in Th2/IL-13, "T22"/IL-22, S100A7 and S100A8, Th1/IFN-gamma, and Th17/IL-17A jointly correlated assessed as change at week 24 compared to baseline of the biomarkers combined z-score expression. Th2/IL-13, T22/IL-22, S100A7 and S100A8, Th1/IFN-gamma, and Th17/IL-17A biomarkers was computed as following. The combined score was obtained by mean z-score expression of all biomarkers, where z-score normalized expression of biomarker X and sample i was obtained by the following formula:
  [Xi - mean(Xall_samples)]/sd(Xall_samples). Change in combined z-score for each patient was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: Baseline and Week 24
Population: data only for those participants who had a biopsy. No participants in placebo group had a biopsy.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 2 | 0
z-score | -0.28 (1.61) |

2. Secondary Outcome: Percentage Change From Baseline in the Severity of Alopecia Tool (SALT)
Description: Percentage change from Baseline in the Severity of Alopecia Tool (SALT) at Week 24.
  SALT score 0-100 with lower score indicating better health outcomes.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 2 | 1
percentage change | 0.49 (33.75) | 0 (0)

3. Secondary Outcome: Number of Patients Achieving 50% or Greater Improvement in Their SALT Score (SALT50)
Description: Number of patients achieving 50% or greater improvement in their SALT score (SALT50) at Week 24, compared to Baseline. SALT score 0-100 with lower score indicating better health outcomes.
Time Frame: Baseline and Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Secondary Outcome: Percentage Change From Baseline in the Alopecia Areata Symptom Impact Scale (AASIS)
Description: Percentage change from baseline in the Alopecia Areata Symptom Impact Scale (AASIS) at Week 24.
  AASIS score 0-130 with lower score indicating better health outcomes.
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 2 | 1
percent change
  baseline | 64 (35.36) | 69 (0)
  week 24 | 57 (52.33) | 50 (0)

5. Secondary Outcome: Percentage Change From Baseline in the Alopecia Areata Quality of Life Questionnaire (AA-QoL)
Description: Percentage change from Baseline in the Alopecia Areata Quality of Life questionnaire (AA-QoL) at Week 24. AA-QoL score 0-100 with higher score indicating better health outcomes.
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 2 | 1
percentage change
  baseline | 59 (14.14) | 47 (0)
  week 24 | 58 (22.63) | 35 (0)

6. Other Pre Specified Outcome: Number of Adverse Events
Description: Side effects to study the safety of tralokinumab in patients with moderate to severe alopecia areata and in patients with concomitant moderate to severe alopecia areata and atopic dermatitis
Time Frame: Week 40
Measure: Number; unit: events
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 15 | 7
events | 8 | 3

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Tralokinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7
Other Adverse Events (participants affected / at risk) | 8/15 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tralokinumab (N=15) | Placebo (N=7)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Upper Respiratory Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypertensive Urgency (Cardiac disorders) | 0 | 1
Corneal Abrasion (Eye disorders) | 1 | 0
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT02684097/Prot_SAP_000.pdf